CLINICAL TRIAL: NCT04592146
Title: POSITIVE: Maintaining and imPrOving the intrinSIc capaciTy Involving Primary Care and caregiVErs
Brief Title: Maintaining and imPrOving the intrinSIc capaciTy Involving Primary Care and caregiVErs
Acronym: POSITIVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Getafe (Other)
Collaborators: Karolinska Institutet (Other); Medical University of Lodz (Other); Universidad Politecnica de Madrid (Other); KTH Royal Institute of Technology (Other); Fundación para la Investigación Biomédica - Hospital Universitario de Getafe (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POSITIVE
Record Dates: First submitted 2020-09-30; First posted 2020-10-19 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2020-10

CONDITIONS: Frailty; Frailty Syndrome; Frail Elderly Syndrome
Keywords: Frailty; Technology; Home monitoring; Older persons
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Multi-centre, non-inferiority, randomized, simple blind and prospective pilot study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Participants randomized into the intervention group will receive care according to the current organizational model in each pilot site (managed by community care). Frailty care will consist in a multicomponent intervention.
  Interventions: Other: Frailty multicomponent intervention
- Intervention group (Experimental): Participants randomized into the intervention group will receive the same intervention as those allocated into the control group, but this intervention will be supported by the POSITIVE technology.Informal caregivers will also receive an app to follow the evolution of the cared person.
  As in the control group, participants allocated into the intervention group will be managed by community care; these professionals will have access to the evolution of the older persons so they can take promote actions in case early deterioration is detected.
  Interventions: Device: Frailty multicomponent intervention supported by POSITIVE; Other: Frailty multicomponent intervention

INTERVENTIONS:
Device: Frailty multicomponent intervention supported by POSITIVE — This technology mainly consists in a home monitoring kit periodically measuring gait speed, involuntary weight loss and power in the lower limb. Furthermore, through a tablet device, other relevant information (e.g. state of mind, activities of daily living-ADLs, etc.) is collected. The same device is used to enhance communication with the clinical team and follow the tailored intervention
  Arms: Intervention group
Other: Frailty multicomponent intervention — This intervention is based on 3 main pillars: medication review (to avoid polypharmacy), tailored nutritional recommendations and a tailored physical activity plan based on the VIVIFRAIL program.

SUMMARY:
The POSITIVE platform offers the possibility of unsupervised monitoring of pre-frailty and frailty status in a community setting, to detect the onset of frailty and to assess its evolution.

The primary objective of the study is to evaluate whether the POSITIVE system improves frailty in at least 1 point in the Fried's Criteria and 5 points in the FTS-5.

This is a multi-centre, non-inferiority, randomized, simple blind and prospective pilot study with a 12-month follow up duration. The study will be carried out in Spain, Sweden and Poland. 150 participants will be randomized into two groups. The control group will receive usual medical care. The intervention group will receive, in addition, the POSITIVE frailty home monitoring and intervention system.

DETAILED DESCRIPTION:
The primary endpoints is to evaluate whether a multimodal intervention supported by the POSITIVE technological ecosystem improves frailty in at least 1 point in Fried's Criteria and 5 points in FTS-5 during a 6-month follow-up period.

This objective will be investigated through a multi-centre, non-inferiority, randomized, simple blind and prospective pilot study with an intervention lasting for 6 months. The study will be carried out in Spain, Sweden and Poland. 150 participants (50 per site) will be randomized into two groups. The control group will receive usual medical care. The intervention group will receive, in addition, the POSITIVE frailty home monitoring and intervention system.

Both groups will be assessed with the same instruments. This assessment will be conducted at baseline (in the beginning of the trial period), at the middle (month 3) and at the end of the intervention (month 6).

A stratified randomization technique will be applied in each of the study groups based on: age group (70-85,> 85), history of cognitive impairment, history of stroke to guarantee the existence of comparable groups. These factors have been significantly associated with frailty and pre-frailty status (stroke OR =3.11 (1.05-9.18), age, per 1-year OR = 1.14 (1.08-1.21); cognitive impairment OR = 8.37 (4.43-15.83)).

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 70.
* Living at home.
* Having a caregiver/relative and/or supervision at home.
* Barthel ≥ 90.
* Meet at least 1 criterion from Fried's Criteria.

Exclusion criteria:

* Inadequate home infrastructure to host the required technology.
* Inability to understand on how to use the POSITIVE system by the participant.
* Diseases that may affect prescription therapy:
* History of alcohol/drugs abuse.
* Living with another participant.
* Participating in other clinical studies.
* Three or more hospitalizations in the last year.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Frailty status 1 | 6 months
  Evaluation of the impact of the technology supported intervention in terms of frailty measured with the Linda Fried's criteria. This test ranges from 0 to 5 (0: robust; 1-2: pre-frailty; +2: frailty).
Frailty status 2 | 6 months
  To evaluate whether a multimodal intervention supported by the POSITIVE technological ecosystem improves frailty in at least 5 points in Frail trait scale (FTS-5) during a 6-month follow-up period. FTS scores between 0-50. 0 is the best value and 50 the worst value.

SECONDARY OUTCOMES:
Frailty trajectories 1 | 6 months
  Trajectories of frailty according to changes in Fried´s phenotype. Fried´s Phenotype scores between 0 and 5. 0 means robust; 1-2 mean pre-frail and 3 or more mean frail
Frailty trajectories 2 | 6 months
  To evaluate whether the POSITIVE system improves frailty transitions in pre-frail and frail participants according to FTS-5.
Physical function 1 | 6 months
  To evaluate whether the POSITIVE system improves participants' physical performance according to the Short Physical Performance Battery (SPPB).SPPB scores between 0-12. 0 is the worst and 12 the best value.
Physical function 2 | 6 months
  To evaluate whether the POSITIVE system improves participants' physical performance according to the Gait Speed test (meters/second)
Basic activities daily living (BADL) | 6 months
  To evaluate the influence of the POSITIVE system in patients' autonomy every day life (basic activities) according to the Barthel Index. Barthel scores between 0-100; 0 is the worst value and 100 the best.
Disability | 6 months
  To evaluate the influence of the POSITIVE system in patients' autonomy every day life (instrumental activities) according to WHO Disability Assessment Schedule (WHODAS 2.0). Score between 0 to 100 (where 0 = no disability; 100 = full disability)
Instrumental activities of daily living (IADL) | 6 months
  To evaluate the influence of the POSITIVE system in patients' autonomy every day life (instrumental activities) according to the Lawton and Brody scale. Lawton and Brody scale scores between 0-10; 0 is the worst and 10 the best value.
Health-related quality of life | 6 months
  To evaluate the influence of the POSITIVE system in the quality of life according to the European Quality of life 5 dimensions-5 levels (EuroQoL 5D-5L). EuroQoL scores between 0-10 and 10 is the worst quality of life.
Cognitive impairment 1 | 6 months
  To evaluate the influence of the POSITIVE system in the cognitive sphere according to the MONTREAL COGNITIVE ASSESSMENT (MoCA test). Scores between 0-30 being 30 the best value.
Cognitive impairment 2 | 6 months
  To evaluate the influence of the POSITIVE system in the cognitive sphere according to the clock drawing test. Score ranges between 0-10. <8 suggests that cognitive impairment (CI)
Affective sphere | 6 months
  To evaluate the influence of the POSITIVE system in the affective sphere according Geriatric Depression Scale (GDS). Each answer indicating depression (bold 'yes' or 'no) counts one point. Scores greater than 5 are indicative of probable depression.
  In the experimental site located in Sweden, the version of this scale will be used.
Caregiver quality of life | 6 months
  To evaluate the influence of the POSITIVE system on the caregiver quality of life according EuroQoL-5D-5L.
To evaluate the usability of the POSITIVE system according to the System Usability Scale (SUS). | 6 months
  SUS ranges from 0 to 100. A SUS score above a 68 would be considered above average and anything below 68 is below average..

CONTACTS AND LOCATIONS:
Overall Officials: Leocadio Rodríguez-Mañas, MD, PhD, Principal Investigator — Hospital Universitario de Getafe; Rodrigo Pérez-Rodríguez, PhD, Principal Investigator — FIB-Hospital Universitario de Getafe
Locations (3):
- Medical University of Lodz, Lodz, Poland
- Fundación para la Investigación Biomédica - Hospital Universitario de Getafe, Getafe, Madrid, Spain
- Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Derived] Terio M, Perez-Rodriguez R, Guevara Guevara T, Valdes-Aragones M, Kornevs M, Bjalevik-Chronan S, Taloyan M, Meijer S, Guidetti S. Preventing frailty with the support of a home-monitoring and communication platform among older adults-a study protocol for a randomised-controlled pilot study in Sweden. Pilot Feasibility Stud. 2022 Aug 23;8(1):190. doi: 10.1186/s40814-022-01147-4. PMID 35999616
- See also: Website to the project site within the EIT-Health website (funding body) European Institute of Innovation & technology — https://eithealth.eu/project/positive/